CLINICAL TRIAL: NCT00453323
Title: A Phase II Study of Weekly Paclitaxel and Capecitabine in Patients With Metastatic or Recurrent Esophageal Cancer
Brief Title: Paclitaxel and Capecitabine in Patients With Metastatic/Recurrence Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Heung Tae Kim, National Cancer Center, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-05-156
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Phase II; Metastatic esophageal cancer; Recurrent esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study arm (Experimental)
  Interventions: Drug: Paclitaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: Paclitaxel — paclitaxel 80mg/m2 iv on day 1 and 8, every 3 weeks
Drug: Capecitabine — capecitabine 900mg/m2 bid po on day 1~14, 1 weeks rest, until disease progression

SUMMARY:
Capecitabine is an orally administered fluoropyrimidine that is converted by 5-FU by thymidine phosphorylase (TP), preferentially in tumor tissues and has demonstrated activity as single agent in patients with gastrointestinal cancer. Up-regulation of TP after taxane treatment in vitro suggested that there may be synergistic effects in combined treatment with taxane and capecitabine. The combination of taxane and capecitabine was reported to be highly active against non-small cell lung cancer, breast cancer, and stomach cancer.

DETAILED DESCRIPTION:
Paclitaxel-80 mg/m2/IV D1 & D8 q 3 weeks Capecitabine-900 mg/m2/PO twice daily Days 1-14 q 3 weeks

Patients receive treatment every 3 weeks till disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed esophageal cancer with histology of squamous carcinoma or adenocarcinoma
2. Clinically diagnosed metastatic or recurrent esophageal cancer according to Sixth Edition of the AJCC Cancer Staging Manual (Appendix V)
3. At least 18 years old
4. Disease status must be that of measurable disease defined as RECIST:Lesions that can be accurately measured in at least one dimension > 10 mm with chest x-ray, spiral CT scan or physical examination
5. ECOG performance status 0-2
6. No prior radiotherapy to measurable lesion(s) but previous surgery and/or chest radiotherapy for the primary lesion is allowed
7. Adequate major organ function including the following:Hematologic function: WBC ≥ 3,500/mm3 or absolute neutrophil count (ANC) ≥ 1,500/mm3, platelet count ≥ 100,000/mm3Hepatic function: bilirubin ≤ 1.5 x UNL , AST/ALT levels ≤ 2.5 x UNLRenal function: serum creatinine ≤ 1.5mg/dL
8. Patients should sign an informed consent
9. If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative hCG test within 7 days prior to the study enrollment.

Exclusion Criteria:

1. MI within preceding 6 months or symptomatic heart disease including unstable angina, congestive heart failure, or uncontrolled arrhythmia
2. Serious concurrent infection or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complication of study therapy
3. Pregnant or nursing women
4. Other malignancy with the past 5 years except adequately treated cutaneous basal cell carcinoma or uterine cervix in situ cancer
5. Psychiatric disorder that would preclude compliance.
6. Major surgery other than biopsy within the past two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-06; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the response rate | the ratio between the number of responders and number of patients assessable for tumor response

SECONDARY OUTCOMES:
To access the toxicity | the first day of the treatment to 30 days after the last dose of study drug
To estimate the time to progression and overall survival | the first day of treatment to the date that disease progression is reported
To evaluate the expression of TP in tumor tissues as a predictive marker for paclitaxel-capecitabine chemotherapy. | before the first treatment
To estimate the overall survival | the first day of the treatment to death date

CONTACTS AND LOCATIONS:
Overall Officials: Heung Tae Kim, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Yun T, Han JY, Lee JS, Choi HL, Kim HY, Nam BH, Kim HT. Phase II study of weekly paclitaxel and capecitabine in patients with metastatic or recurrent esophageal squamous cell carcinoma. BMC Cancer. 2011 Sep 2;11:385. doi: 10.1186/1471-2407-11-385. PMID 21888637